CLINICAL TRIAL: NCT02426385
Title: Comparison of Viusal Outcomes After Implantation of the POD 26% FineVision
Brief Title: Comparison of Viusal Outcomes After Implantation of the POD 26% FineVision Toric (PhysIOL) and POD 26% Toric (PhysIOL)
Status: Withdrawn | Type: Observational
Why Stopped: lack of suitable patients
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TaneriPODAYFT/PODAYT
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1POD26PFT: Patients implanted with the POD 26% FineVision Toric
  Interventions: Device: FineVision Toric
- 2POD26PT: Patients implanted with the POD 26% Toric

INTERVENTIONS:
Device: FineVision Toric — Posterior chamber IOL which consists in a small plastic lens with plastic side struts, called haptics, to hold the lens in place within the capsular bag inside the eye
  Groups: 1POD26PFT

SUMMARY:
The study is an observational non-randomised controlled study comparing the visual acuity after implantation of the POD 26% FINEVISION TORIC with respect to the POD 26% TORIC

DETAILED DESCRIPTION:
The study is an observational non-randomised controlled study comparing the visual acuity after implantation of the POD 26% FINEVISION TORIC with respect to the POD 26% TORIC This study includes both eyes of 24 patients implanted with the POD 26%FineVision Toric (group 1: 12 patients) and the POD 26% Toric (group 2: 12 patients) .

The study primary goal is to compare the near visual acuity in both groups. Distance and intermediate visual acuities, defocus curve, refraction and straylight will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 50 years old
* Regular corneal astigmatism >1.0 dioptres by IOL Master (regularity determined by the topography of the keratometry).
* Regular corneal astigmatism <2.5 dioptres by IOL Master (regularity determined by the topography of the keratometry).
* Group 1: patients after cataract surgery with Fine Vision toric implanted in both eyes
* Group 2: patients after cataract surgery with Ankoris implanted in both eyes
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

• - Irregular astigmatism

* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalitis (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* IOL spherical equivalent power lower than 10 D or greater than 30D
* Complicated surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pseudophakic patients implanted with one of the two IOLs
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The visual acuity at near of the POD 26% FINEVISION TORIC with respect to the POD 26% TORIC is improved of at least LogMAR 0.2. | 3 months

SECONDARY OUTCOMES:
The secondary objective is to measure far and intermediate visual acuity, the refraction, centration, rotational stability and to determine the amount of photic phenomena for both IOLs: POD 26% FINEVISION TORIC and POD 26% TORIC. | 3 months